CLINICAL TRIAL: NCT06579066
Title: The Effect of Probiotics Versus Activated Charcoal in the Management of Chronic Kidney Disease Patients Suffering From Uremic Pruritus.
Brief Title: The Effect of Probiotics vs Activated Charcoal in the Management of CKD Patients Suffering From Uremic Pruritus.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aliaa Mohamed Ashraf Mohamed HaGr, Dr Aliaa Mohamed, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uremic Pruitus
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease; Uremic Pruritus
Keywords: Probiotics; Activated Charcoal; uremic pruritus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anthrax | interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: One hundred twenty three patients who will fit the inclusion criteria will be randomly divided into 3 groups:
  Group 1 (Probiotics group): 41 Patients will administer Linex®(one capsule daily) orally along with the standard care of therapy for duration of 4 weeks.
  Group 2 (activated charcoal): 41 Patients will administer Charclone® 1000MG Tab (Tablet three times daily) orally along with the standard care of therapy for duration of 4 weeks.
  Patients will take activated charcoal dose at least 2 hours before taking other drugs.
  Group 3 (Control group) : 41 Patients will administer standard care of therapy alone (fexofenadine) TELFAST®120mg tablet once daily
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- probiotics (Experimental): Patients will administer Linex ® capsule orally along with the standard care of therapy for duration of 4 weeks.
  Dose: Capsule once daily
  Interventions: Drug: Probiotic Blend Capsule
- activated charcoal (Experimental): Patients will administer Charclone® 1000mg tab orally along with the standard care of therapy for duration of 4 weeks.
  Dose: Tablet three times daily.
  Interventions: Drug: Activated Charcoal
- Control (No Intervention): Patients will administer standard care of therapy alone Telfast®120mg tablet for duration of 4 weeks.. Dose: Tablet once daily

INTERVENTIONS:
Drug: Probiotic Blend Capsule — Patients will administer (probiotics) Linex® one capsule daily orally along with the standard care of therapy for duration of 4 weeks.
  Other Names: linex®
  Arms: probiotics
Drug: Activated Charcoal — Patients will administer (activated charcoal) Charclone® 1000MG Tablet three times daily orally along with the standard care of therapy for duration of 4 weeks.
  Other Names: Charclone®
  Arms: activated charcoal

SUMMARY:
This study aims to evaluate the efficacy and safety of probiotics versus activated charcoal in management of chronic kidney disease patients suffering from uremic pruritus.

Patient data collection

Demographic data:The following data will be collected from the patient records; including age, sex, weight, height.

History Taking :Including patient's medical history, past surgical history, family medical history, and medications the patient is taking or may have recently stopped taking.

A patient's medical history may also include information about allergies, etiology of uremic pruritus.

Laboratory examinations:The following laboratory data to be measured at baseline and after the duration of treatment (4 weeks)

1. Serum levels of indoxyl sulfate (IS)
2. Kidney Function tests: BUN, Creatinine
3. Electrolytes test: sodium, potassium, chloride ,ionized calcium, phosphorus

Dermatological examination: Base on

1. measure Visual Analoge Scale Score(VAS).
2. measure Dermatology life quality index (DLQI).

DETAILED DESCRIPTION:
Chronic kidney disease-associated pruritus (CKD-aP) , also called uremic pruritus (UP) is a critical problem defined as un pleasant sensation that desire to itch and scratch experienced by people with chronic kidney disease (CKD) patients . Pruritus is the most common skin symptoms related with uremia and has a major clinical effect being associated strongly with poor quality of life , impaired sleep and increased mortality, so it's important to explore an efficient treatment option for it. Although the pathogenesis of pruritus remains largely unclear, it is demonstrated that pruritus is mainly ascribed to the retention of uremic solutes.

Gut microbiome has gained attention and is increasingly noted to play a significant role in a number of disorders including CKD. Patients with CKD can be characterized with lower bacterial richness and diversity. Like the gut, human skin has its own microbiome. Recent study showed that CKD patients with pruritus had a different bacterial community comparing to those without pruritus indicating that altered skin microbiome associated with pruritus in patients with CKD and also with accumulation of uremic toxins in skin. So, the skin microbiome plays a potential role in regulating the skin symptoms in CKD patients. Therefore, these findings might be useful for making probiotics supplements to relieve patient's skin symptoms or renal damage.

Indoxyl sulfate (IS) is one of the most potent protein bound uremic toxins derived from the gut microbes. IS is generated by bacterial metabolism of trptophan to indole. The serum IS was significantly elevated in patients with CKD associated pruritus. Moreover, High serum IS concentration has a strong relationship with pruritus severity and a negative impact on quality of life. Therefore, IS may represent a potential therapeutic target to reduce the pruritus severity.

To decrease serum IS levels either decrease IS production by using probiotic supplementation or decrease IS intestinal absorption by addition of activated charcoal as an adsorbent agent has been evaluated in uremic patients.

Probiotics are defined as live microorganisms that consumed in adequate amounts; confer a health effect on the host. Probiotics supplement regulating the immune system and improving the skin barrier. Probiotics work by competing with pathogenic organisms for nutrients, which prevent the growth of harmful bacteria. So, probiotics has a key role in improving the microbiota.Several clinical trials are being carried out on the efficacy of probiotics for the treatment of many skin problems. Some trials also showed that probiotics has a role in reducing of protein bound uremic toxin such indoxyl sulfate (IS).We hope that this study forms a contribution to promoting probiotics as a novel therapeutic approach for the treatment of uremic pruritus.

Activated charcoal is a powerful, intestinal adsorbent within the gastrointestinal (GI) tract, effectively trapping various chemicals. These captured substances are then retained within the charcoal matrix, preventing or reducing their absorption into the blood stream. Activated charcoal has been found to effectively eliminate urea and other uremic toxin such as indoxyl sulfate due to its ability to bind with IS and expelling it through feces. It's also showed that the usage of activated charcoal resulted in decreasing pruritus severity and improving the quality of life of patients without serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with uremic pruritus aged from 18 years and older will be enrolled in the study.

Exclusion Criteria:

1. Patients with psoriasis, atopic dermatitis or any other condition that can justify pruritus.
2. Patient undergoing dialysis.
3. Patients with known allergy to Activated charcoal or probiotics supplements.
4. Patients who are non-compliant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in serum Indoxyl sulfate (IS) level | Four weeks
  IS is one of the most potent protein bound uremic toxins . mesasuring serum indoxyl sulfate level at baseline and after a 4 weeks trial period by using ELISA kits.
Change in visual Analog scale (VAS) score. | Four weeks
  A 10 cm horizontal line marked from zero (no pruritus) to 10 (worst possible pruritus). The pruritus will be assessed subjectively and scored at baseline and after a 4 weeks trial period .
Change in Dermatology life quality index (DLQI) | Four weeks
  10-Item questionnaire aiming to measure how much skin problem has affected on QOL . mesasuring DLQI at baseline and after a 4 weeks trial period .

SECONDARY OUTCOMES:
Evaluation of the safety of probiotics supplementation and activated charcoal in patients with uremic pruritus. | Four weeks
  by monitor any adverse effects that may occur throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Mohamed, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akl EM, El-Eraki JM, Elfallah AA, Mohamed NH, Maher AM, Mansour AE, Abdelsalam OH. Does Indoxyl Sulfate Have a Role in Uremic Pruritus? A Laboratory and Interventional Study. J Cutan Med Surg. 2024 Jan-Feb;28(1):44-50. doi: 10.1177/12034754231220935. Epub 2023 Dec 29. PMID 38156627
- [Background] Kim SH, Jhee JH, Choi HY, Lee SH, Shin SK, Lee SY, Yang DH, Yi JH, Han SW, Jo YI, Park HC. New oral spherical carbon adsorbent effectively reduces serum indoxyl sulfate levels in moderate to advanced chronic kidney disease patients: a multicenter, prospective, open-label study. BMC Nephrol. 2020 Jul 31;21(1):317. doi: 10.1186/s12882-020-01971-x. PMID 32736531
- [Background] Szanto M, Dozsa A, Antal D, Szabo K, Kemeny L, Bai P. Targeting the gut-skin axis-Probiotics as new tools for skin disorder management? Exp Dermatol. 2019 Nov;28(11):1210-1218. doi: 10.1111/exd.14016. Epub 2019 Aug 28. PMID 31386766